CLINICAL TRIAL: NCT04707508
Title: Investigating the Effect of Renin-Angiotensin System Inhibitors in Addition to Standard Antidiabetic Therapy on Glycemic Control in Patients With Type 2 Diabetes Mellitus: A Prospective Open-label Study
Brief Title: Effect of Adding Renin-Angiotensin System Inhibitors to Standard Antidiabetic Therapy on Glycemic Control in Patients With Type 2 Diabetes Ellitus
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nantou Christian Hospital (Other)
Responsible Party: Principal Investigator, Po-Chung Cheng, Director, Division of endocrine and metabolic diseases, Nantou Christian Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Y_106_0298
Record Dates: First submitted 2021-01-11; First posted 2021-01-13 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2021-01

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Valsartan; Metformin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Valsartan and metformin (Experimental)
  Interventions: Drug: Valsartan 80 mg and metformin
- Metformin only (Active Comparator)
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Valsartan 80 mg and metformin — Valsartan 80 mg once daily in addition to metformin monotherapy
  Arms: Valsartan and metformin
Drug: Metformin — Metformin monotherapy
  Arms: Metformin only

SUMMARY:
Type 2 diabetes mellitus (T2DM) is a progressive metabolic disorder in which a substantial number of patients cannot attain treatment target despite antidiabetic drugs. The renin-angiotensin system (RAS) has recently been implicated in the development of insulin resistance and impaired glucose metabolism. This study investigates the effect of adding RAS inhibitors to standard antidiabetic therapy in patients with T2DM. The primary outcome measure is the change in serum glycosylated hemoglobin A1c after 24 weeks of treatment. Secondary outcomes measures include changes in plasma lipid profile and blood pressure after treatment.

ELIGIBILITY:
Inclusion Criteria:

* adults over 21 years of age
* clinically diagnosed type 2 diabetes mellitus
* recipients of metformin monotherapy
* compliance with prescriptions and dietary intervention

Exclusion Criteria:

* recipients of any second-line antidiabetic drug in addition to metformin
* recipients of any antihypertensive medication before study enrollment
* hemoglobin disorders
* chronic kidney disease
* thyroid dysfunction

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 203 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2019-11-29 (Actual)

PRIMARY OUTCOMES:
Serum glycosylated hemoglobin A1c | 24 weeks
  Change in serum glycosylated hemoglobin A1c of the participants

SECONDARY OUTCOMES:
Plasma lipid fractions | 24 weeks
  Change in plasma triglycerides, high-density lipoprotein cholesterol, low-density lipoprotein cholesterol
Blood pressure | 24 weeks
  Change in systolic blood pressure and diastolic blood pressure

CONTACTS AND LOCATIONS:
Overall Officials: Po-Chung Cheng, MD, Principal Investigator — Nantou Christian Hospital
Locations (1):
- Nantou Christian Hospital, Nantou City, Nantou County, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khan MAB, Hashim MJ, King JK, Govender RD, Mustafa H, Al Kaabi J. Epidemiology of Type 2 Diabetes - Global Burden of Disease and Forecasted Trends. J Epidemiol Glob Health. 2020 Mar;10(1):107-111. doi: 10.2991/jegh.k.191028.001. PMID 32175717
- [Background] Nehme A, Zouein FA, Zayeri ZD, Zibara K. An Update on the Tissue Renin Angiotensin System and Its Role in Physiology and Pathology. J Cardiovasc Dev Dis. 2019 Mar 29;6(2):14. doi: 10.3390/jcdd6020014. PMID 30934934
- [Background] Joseph JJ, Echouffo Tcheugui JB, Effoe VS, Hsueh WA, Allison MA, Golden SH. Renin-Angiotensin-Aldosterone System, Glucose Metabolism and Incident Type 2 Diabetes Mellitus: MESA. J Am Heart Assoc. 2018 Sep 4;7(17):e009890. doi: 10.1161/JAHA.118.009890. PMID 30371168
- [Background] Das UN. Renin-angiotensin-aldosterone system in insulin resistance and metabolic syndrome. J Transl Int Med. 2016 Jun 1;4(2):66-72. doi: 10.1515/jtim-2016-0022. Epub 2016 Jul 7. PMID 28191524
- [Background] Mor A, Aizman E, George J, Kloog Y. Ras inhibition induces insulin sensitivity and glucose uptake. PLoS One. 2011;6(6):e21712. doi: 10.1371/journal.pone.0021712. Epub 2011 Jun 29. PMID 21738773